CLINICAL TRIAL: NCT02333916
Title: Effects of Short-term Overfeeding With or Without Exercise on 24-hour Fat Oxidation and Fat Balance Before and After 10 Weeks of Training - The FeedEX Study
Brief Title: Effect of Exercise and Training on Fat Oxidation During Overfeeding - the FeedEX Study
Acronym: FeedEX
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment target could not be met
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL47945.068.14
Record Dates: First submitted 2014-12-30; First posted 2015-01-07 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-04

CONDITIONS: Overfeeding and Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overfeeding + exercise pre/post training (Experimental): overfeeding + exercise pre-training: day1 energy balance; day2 and day3: energy intake equals 1.25 times day 2 and day 3 energy expenditure respectively, no exercise; day4: 3 cycling bouts to expend 0.25 times day3 energy expenditure + energy intake equals 1.25 times day4 energy expenditure - before training period.
  fitness training: 10-week training period (3 times per week at a gym, 30-45 minutes cardio training and 15-30 minutes strength training).
  overfeeding + exercise post-training: day1 energy balance; day2 and day3: energy intake equals 1.25 times day 2 and day 3 energy expenditure respectively, no exercise; day4: 3 cycling bouts to expend 0.25 times day3 energy expenditure + energy intake equals 1.25 times day4 energy expenditure - after training period.
  Interventions: Other: overfeeding + exercise pre-training; Behavioral: fitness training; Other: overfeeding + exercise post-training

INTERVENTIONS:
Other: overfeeding + exercise pre-training
Behavioral: fitness training
Other: overfeeding + exercise post-training

SUMMARY:
Rationale: Body weight is not well regulated in all individuals. In an obesogenic environment, where overeating is common, some individuals are more prone to weight gain and therefore overweight than others. Yet, the reasons behind this are unclear. "Resistant" individuals often have higher physical activity levels (PALs). It seems that - at higher levels of physical activity and therefore energy expenditure - satiety signals are more precisely regulated, making one better at matching energy intake with expenditure. In other words, active people may not overeat where sedentary people would. However, this does not explain the differences in weight gain observed when subjects all have to overeat (imposed overfeeding). It could be that active people are better able to cope metabolically with the extra calories because of already higher levels of carbohydrate and fat oxidation compared to their inactive counterparts.

Objectives: 1/ To study the effects of overfeeding (normal diet composition) on substrate balance and oxidation and more specifically fat balance and oxidation; 2/ to study the effects of exercise and training on fat oxidation during overfeeding (normal diet composition).

Study design: This controlled intervention study will follow a cross-over design. Each subject will spend 5 nights and 4 days in a respiration chamber on two occasions, separated by a 10-week training period.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians
* Male
* Healthy
* 18-30 years
* BMI 21-27.5 kg.m-2
* Sedentary lifestyle: the following serve as (non-strict) guidelines: "Low category of activity" according to the short version of the International Physical Activity Questionnaire (IPAQ); VO2max (ml.kg-1.min-1) below: 45 - AGE (yrs) / 3 corresponding to a fitness category below "fair" (i.e. "poor" or "very poor") as defined by Schvartz and Reibold. For example for an 18 year-old male, VO2max below 39 ml.kg-1.min-1.
* Stable body weight (<5% change in the last 6 months)

Exclusion Criteria:

* Following a (weight-loss) diet
* Using medications
* Smoking
* Consuming more than 3 units of alcohol per day
* Diagnosed with any chronic diseases known to affect energy metabolism (intake/expenditure) such as diabetes, cardiovascular disease, cancer, or thyroid disease.
* Trained or regularly physically active (according to the IPAQ)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour fat balance with overfeeding after training | Baseline and 3 months
  Day3 24-hour fat balance (calculated as the difference between metabolisable fat intake and fat oxidation measured by indirect calorimetry in respiration chamber) after training compared to baseline (=before training)
Change in 24-hour fat balance with overfeeding and exercise after training | Baseline and 3 months
  Day4 24-hour fat balance (calculated as the difference between metabolisable fat intake and fat oxidation measured by indirect calorimetry in respiration chamber) after training compared to baseline (=before training)

SECONDARY OUTCOMES:
Change in 24-hour fat oxidation with overfeeding and exercise in inactive men | Day 3 and day 4 (baseline stay in respiration chamber)
  Fat oxidation measured by indirect calorimetry in respiration chamber on day 4 compared to day 3 at baseline
Change in 24-hour carbohydrate oxidation with overfeeding and exercise in inactive men | Day 3 and day 4 (baseline stay in respiration chamber)
  Carbohydrate oxidation measured by indirect calorimetry in respiration chamber on day 4 compared to day 3 at baseline
Change in 24-hour fat balance with overfeeding and exercise in inactive men | Day 3 and day 4 (baseline stay in respiration chamber)
  Fat balance (calculated as the difference between metabolisable fat intake and fat oxidation) on day 4 compared to day 3 at baseline
Change in 24-hour fat oxidation with overfeeding and exercise in active men | Day 3 and day 4 (stay in respiration chamber at 3 months)
  Fat oxidation measured by indirect calorimetry in respiration chamber on day 4 compared to day 3 after the training period
Change in 24-hour carbohydrate oxidation with overfeeding and exercise in active men | Day 3 and day 4 (stay in respiration chamber at 3 months)
  Carbohydrate oxidation measured by indirect calorimetry in respiration chamber on day 4 compared to day 3 after the training period
Change in 24-hour fat balance with overfeeding and exercise in active men | Day 3 and day 4 (stay in respiration chamber at 3 months)
  Fat balance (calculated as the difference between metabolisable fat intake and fat oxidation) on day 4 compared to day 3 after the training period
Change in 24-hour carbohydrate oxidation with overfeeding after training | Baseline and 3 months
  Day3 24-hour carbohydrate oxidation measured by indirect calorimetry in respiration chamber after training compared to baseline (=before training)
Change in 24-hour carbohydrate oxidation with overfeeding and exercise after training | Baseline and 3 months
  Day4 24-hour carbohydrate oxidation measured by indirect calorimetry in respiration chamber after training compared to baseline (=before training)
Change in fat oxidation after training assessed in energy balance | Baseline and 3 months
Change in carbohydrate oxidation after training assessed in energy balance | Baseline and 3 months
Energy expenditure with overfeeding in inactive men | 4 days at baseline
  Energy expenditure measured by indirect calorimetry during a 4-day stay in respiration chamber, with overfeeding on days 2 to 4.
Energy expenditure with overfeeding in active men | 4 days at 3 months
  Energy expenditure measured by indirect calorimetry during a 4-day stay in respiration chamber, with overfeeding on days 2 to 4, after a 10-week fitness training.
Insulin sensitivity | Baseline, 2 weeks (pre-training), 3 months (post-training)
  Based on glucose and insulin plasma concentrations from oral glucose tolerance test, where blood is collected in fasted state at t=0, 30, 60, 90 and 120min after a glucose drink is ingested)
adipocyte size | Baseline, 2 weeks (pre-training), 3 months (post-training)
  Fat biopsy taken these time points
Genes involved in lipid metabolism | Baseline, 2 weeks (pre-training), 3 months (post-training)
  Using fat biopsies: analysis of genes involved in the lipolytic pathway [ATGL (PNPLA2), HSL (S660/565/563), CGI-58, G0S2, PLIN1, AQP7, GK], in insulin signaling/glucose metabolism [GLUT4, IRS1/IRS2, AKT, pAKT (S473), pIRS1 (S1101)], in fatty acid metabolism [CD36, FABP4 (aP2), FASN, CPT1a/1b, CPT2, ACADL/ACADVL/ACADS/ACADM, ACOX1, OXPHOS (complex I-V), PPAR(α/βδ/γ), PGC1a, PGC1b, SIRT1, AMPK (pAMPK)], and in DAG/ceramide metabolism [DGAT 1/2, GPAT1/GPAM, PLC, SPTLC1 and SPTLC2, CERK, ASAH1 and ASAH2
Change in body composition | Baseline and 3 months
  Measured using body weight, underwater weighing and deuterium dilution, before and after the fitness training
Change in cardiorespiratory fitness | Baseline, after 6-7 weeks of training and 3 months
  Cardiorespiratory fitness estimated as the maximal oxygen uptake (VO2max) assessed using an incremental test on a bicycle ergometer
Change in energy expenditure in free-living conditions | Baseline and 3 months
  Energy expenditure measured over 14 days using doubly-labeled water and two accelerometers (TracmorD and Actigraph GT3X)
Validity of Actigraph GT3X accelerometer | Two 14-day periods (baseline and 3 months)
  The Actigraph GT3X accelerometer is worn by each subject twice for 14 days and will be validated against the doubly labeled water technique and compared to the tracmorD accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Wim Saris, MD, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Schokker DF, Visscher TL, Nooyens AC, van Baak MA, Seidell JC. Prevalence of overweight and obesity in the Netherlands. Obes Rev. 2007 Mar;8(2):101-8. doi: 10.1111/j.1467-789X.2006.00273.x. PMID 17300276
- [Background] Bouchard C, Tremblay A, Despres JP, Nadeau A, Lupien PJ, Theriault G, Dussault J, Moorjani S, Pinault S, Fournier G. The response to long-term overfeeding in identical twins. N Engl J Med. 1990 May 24;322(21):1477-82. doi: 10.1056/NEJM199005243222101. PMID 2336074
- [Background] Diaz EO, Prentice AM, Goldberg GR, Murgatroyd PR, Coward WA. Metabolic response to experimental overfeeding in lean and overweight healthy volunteers. Am J Clin Nutr. 1992 Oct;56(4):641-55. doi: 10.1093/ajcn/56.4.641. PMID 1414963
- [Background] Joosen AM, Bakker AH, Westerterp KR. Metabolic efficiency and energy expenditure during short-term overfeeding. Physiol Behav. 2005 Aug 7;85(5):593-7. doi: 10.1016/j.physbeh.2005.06.006. PMID 16039676
- [Background] Lammert O, Grunnet N, Faber P, Bjornsbo KS, Dich J, Larsen LO, Neese RA, Hellerstein MK, Quistorff B. Effects of isoenergetic overfeeding of either carbohydrate or fat in young men. Br J Nutr. 2000 Aug;84(2):233-45. PMID 11029975
- [Background] Levine JA, Eberhardt NL, Jensen MD. Role of nonexercise activity thermogenesis in resistance to fat gain in humans. Science. 1999 Jan 8;283(5399):212-4. doi: 10.1126/science.283.5399.212. PMID 9880251
- [Background] Norgan NG, Durnin JV. The effect of 6 weeks of overfeeding on the body weight, body composition, and energy metabolism of young men. Am J Clin Nutr. 1980 May;33(5):978-88. doi: 10.1093/ajcn/33.5.978. PMID 7369169
- [Background] Joosen AM, Bakker AH, Zorenc AH, Kersten S, Schrauwen P, Westerterp KR. PPARgamma activity in subcutaneous abdominal fat tissue and fat mass gain during short-term overfeeding. Int J Obes (Lond). 2006 Feb;30(2):302-7. doi: 10.1038/sj.ijo.0803146. PMID 16247507
- [Background] MAYER J, ROY P, MITRA KP. Relation between caloric intake, body weight, and physical work: studies in an industrial male population in West Bengal. Am J Clin Nutr. 1956 Mar-Apr;4(2):169-75. doi: 10.1093/ajcn/4.2.169. No abstract available. PMID 13302165
- [Background] Hill JO, Wyatt HR, Peters JC. Energy balance and obesity. Circulation. 2012 Jul 3;126(1):126-32. doi: 10.1161/CIRCULATIONAHA.111.087213. PMID 22753534
- [Background] Horton TJ, Drougas H, Brachey A, Reed GW, Peters JC, Hill JO. Fat and carbohydrate overfeeding in humans: different effects on energy storage. Am J Clin Nutr. 1995 Jul;62(1):19-29. doi: 10.1093/ajcn/62.1.19. PMID 7598063
- [Background] Jebb SA, Prentice AM, Goldberg GR, Murgatroyd PR, Black AE, Coward WA. Changes in macronutrient balance during over- and underfeeding assessed by 12-d continuous whole-body calorimetry. Am J Clin Nutr. 1996 Sep;64(3):259-66. doi: 10.1093/ajcn/64.3.259. PMID 8780332
- [Background] Blaak EE, Hul G, Verdich C, Stich V, Martinez A, Petersen M, Feskens EF, Patel K, Oppert JM, Barbe P, Toubro S, Anderson I, Polak J, Astrup A, Macdonald IA, Langin D, Holst C, Sorensen TI, Saris WH. Fat oxidation before and after a high fat load in the obese insulin-resistant state. J Clin Endocrinol Metab. 2006 Apr;91(4):1462-9. doi: 10.1210/jc.2005-1598. Epub 2006 Jan 31. PMID 16449343
- [Background] Blair SN, Brodney S. Effects of physical inactivity and obesity on morbidity and mortality: current evidence and research issues. Med Sci Sports Exerc. 1999 Nov;31(11 Suppl):S646-62. doi: 10.1097/00005768-199911001-00025. PMID 10593541
- [Background] Knudsen SH, Hansen LS, Pedersen M, Dejgaard T, Hansen J, Hall GV, Thomsen C, Solomon TP, Pedersen BK, Krogh-Madsen R. Changes in insulin sensitivity precede changes in body composition during 14 days of step reduction combined with overfeeding in healthy young men. J Appl Physiol (1985). 2012 Jul;113(1):7-15. doi: 10.1152/japplphysiol.00189.2011. Epub 2012 May 3. PMID 22556394
- [Background] Hagobian TA, Braun B. Interactions between energy surplus and short-term exercise on glucose and insulin responses in healthy people with induced, mild insulin insensitivity. Metabolism. 2006 Mar;55(3):402-8. doi: 10.1016/j.metabol.2005.09.017. PMID 16483886
- [Background] Walhin JP, Richardson JD, Betts JA, Thompson D. Exercise counteracts the effects of short-term overfeeding and reduced physical activity independent of energy imbalance in healthy young men. J Physiol. 2013 Dec 15;591(24):6231-43. doi: 10.1113/jphysiol.2013.262709. Epub 2013 Oct 28. PMID 24167223
- [Background] Speakman JR. The history and theory of the doubly labeled water technique. Am J Clin Nutr. 1998 Oct;68(4):932S-938S. doi: 10.1093/ajcn/68.4.932S. PMID 9771875
- [Background] Plasqui G, Joosen AM, Kester AD, Goris AH, Westerterp KR. Measuring free-living energy expenditure and physical activity with triaxial accelerometry. Obes Res. 2005 Aug;13(8):1363-9. doi: 10.1038/oby.2005.165. PMID 16129718
- See also: Related Info — http://www.who.int/mediacentre/factsheets/fs311/en/.
- See also: Related Info — http://www.euro.who.int/en/health-topics/noncommunicable-diseases/obesity/data-and-statistics.